CLINICAL TRIAL: NCT03011203
Title: Acute Nutritional Ketosis and Exercise in Glycogen Storage Disease Type IIIa
Brief Title: Acute Nutritional Ketosis in GSD IIIa
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Medical Center Groningen (Other)
Collaborators: University of the Faroe Islands (Other); University of Oxford (Other); Stichting Stofwisselkracht (Unknown); Stichting Metakids (Unknown)
Responsible Party: Principal Investigator, Terry G.J. Derks, MD, PhD, Pediatrician consultant metabolic medicine, University Medical Center Groningen
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Other
Other Study IDs: NL59081.042.16
Record Dates: First submitted 2016-12-22; First posted 2017-01-05 (Estimated); Last update posted 2018-05-01 (Actual); Status verified 2018-04

CONDITIONS: Glycogen Storage Disease IIIA
Keywords: glycogen storage disease type IIIa; exercise; ketone esters; magnetic resonance spectroscopy
MeSH Terms: conditions — Glycogen Storage Disease IIIA; Motor Activity | interventions — Exercise

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Ketone-ester drink (Experimental): Oral intake - physical exercise
  Interventions: Other: physical exercise
- Carbohydrate drink (Active Comparator): Oral intake - physical exercise
  Interventions: Other: physical exercise

INTERVENTIONS:
Other: physical exercise — In session II and III participants will perform an exercise test on a bicycle inside and outside the MR scanner.

SUMMARY:
The investigators will study if acute nutritional ketosis in adult GSD IIIa patients can boost muscle mitochondrial function in vivo.

DETAILED DESCRIPTION:
Glycogen Storage Disease type IIIa (GSD IIIa) is an inborn error of carbohydrate metabolism caused by impaired glycogen debranching enzyme (GDE) activity. The ageing GSD IIIa cohort shows that muscle involvement -despite dietary management- is a common disabling phenotype in adulthood. Currently, no specific therapy has been established for muscle problems in adult GSD IIIa patients.

However, it could be hypothesized that nutritional ketosis (NK) will be highly beneficial to patients. Amongst others, ketone bodies could take on the role of primary energy source in exercising muscle. Recently, acute NK in exercise was studied in humans. NK was found to enhance muscle mitochondrial function in athletes.

The investigators will study if acute NK in adult GSD IIIa patients can boost muscle mitochondrial function in vivo.

ELIGIBILITY:
Inclusion Criteria:

* GSD III confirmed with enzyme assay and/or AGL mutation analysis and GSD IIIa further specified as deficient debranching enzyme activity in muscle or clinical and/or biochemical signs of cardiac and/or skeletal muscular involvement.

Exclusion Criteria:

* contraindications for MRI studies (assessed by standardised questionnaire)
* inability to perform bicycle exercise.
* intercurrent illness which may influence exercise tolerance (anemia, musculoskeletal injury, or other undiagnosed illness under investigation).
* known coronary artery disease, positive history for angina or cardiomyopathy.
* insulin-dependent diabetes mellitus.
* loss of, or an inability to give informed consent.
* pregnancy or current breastfeeding.
* any other cause which in the opinion of the investigators, may affect the participant's ability to participate in the study

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2017-02-10 (Actual); Primary Completion 2018-03-23 (Actual); Study Completion 2018-03-23 (Actual)

PRIMARY OUTCOMES:
Description of in vivo energy and proton balance during exercise in MR scanner with and without ketone ester drink: steady-state intramuscular levels of glycogen, Pi, PCr and pH and kinetic rate constant of metabolic recovery. | 10 minutes; during in-magnet exercise test of session II and III.

SECONDARY OUTCOMES:
time of individual desired workload | through completion of the maximum exercise test (of approximately 12 minutes) during study session I.
  #minutes
completion of supine bicycling bout at desired workload in scanner | 10 min
  (yes/no; if no, #minutes)
Muscle ultrasound density of the biceps, quadriceps, calf (gastrocnemius and/or soleus) and tibialis anterior muscles. | Together with the muscle force examination this assessment will take 1.5 hour.
  Will be performed during study session I by a neurologist.
Muscle force unilateral | Together with the muscle ultrasound this assessment will take 1.5 hour.
  Will be performed during study session I by a neurologist.
Subjective fatigue and muscle ache score | after each exercise bout and 24 hours after exercise
  scale 0-10
International Physical Activity Questionnaire | This questionnaire will take 10 minutes to fill out. Participants will be asked to fill out the questionnaire one week before study session II and III
Structural muscle parameters: fat infiltration. | During the in-magnet exercise test of 10 minutes during session II and III
Change in blood glucose levels | Up to 7 samples will be taken during the 25 minutes exercise test (session II and III).
  #1 and #2 at baseline, #3 after 10 min, #4 after 15 minutes, #5 at the start of bicycle exercise test inside scanner, #6 after 10 minutes of in-magnet exercise and #7 three hours post-exercise inside scanner.
Blood ketones level (β-hydroxybutyrate, acetoacetate). | Up to 7 samples will be taken during the 25 minutes exercise test (session II and III).
  #1 and #2 at baseline, #3 after 10 min, #4 after 15 minutes, #5 at the start of bicycle exercise test inside scanner, #6 after 10 minutes of in-magnet exercise and #7 three hours post-exercise inside scanner.
Change of blood pH | Up to 7 samples will be taken during the 25 minutes exercise test (session II and III).
  #1 and #2 at baseline, #3 after 10 min, #4 after 15 minutes, #5 at the start of bicycle exercise test inside scanner, #6 after 10 minutes of in-magnet exercise and #7 three hours post-exercise inside scanner.
Blood levels of free fatty acids | Up to 7 samples will be taken during the 25 minutes exercise test (session II and III).
  #1 and #2 at baseline, #3 after 10 min, #4 after 15 minutes, #5 at the start of bicycle exercise test inside scanner, #6 after 10 minutes of in-magnet exercise and #7 three hours post-exercise inside scanner.
Blood levels of insulin | Up to 7 samples will be taken during the 25 minutes exercise test (session II and III).
  #1 and #2 at baseline, #3 after 10 min, #4 after 15 minutes, #5 at the start of bicycle exercise test inside scanner, #6 after 10 minutes of in-magnet exercise and #7 three hours post-exercise inside scanner.
Blood levels of creatine kinase | Up to 7 samples will be taken during the 25 minutes exercise test (session II and III).
  #1 and #2 at baseline, #3 after 10 min, #4 after 15 minutes, #5 at the start of bicycle exercise test inside scanner, #6 after 10 minutes of in-magnet exercise and #7 three hours post-exercise inside scanner.
Blood levels of ammonia | Up to 7 samples will be taken during the 25 minutes exercise test (session II and III).
  #1 and #2 at baseline, #3 after 10 min, #4 after 15 minutes, #5 at the start of bicycle exercise test inside scanner, #6 after 10 minutes of in-magnet exercise and #7 three hours post-exercise inside scanner.
Blood levels of NT-proBNP | Up to 7 samples will be taken during the 25 minutes exercise test (session II and III).
  #1 and #2 at baseline, #3 after 10 min, #4 after 15 minutes, #5 at the start of bicycle exercise test inside scanner, #6 after 10 minutes of in-magnet exercise and #7 three hours post-exercise inside scanner.
Blood levels of lactate | Up to 7 samples will be taken during the 25 minutes exercise test (session II and III).
  #1 and #2 at baseline, #3 after 10 min, #4 after 15 minutes, #5 at the start of bicycle exercise test inside scanner, #6 after 10 minutes of in-magnet exercise and #7 three hours post-exercise inside scanner.
Change of urine levels of myoglobin, ketones, tetraglucoside | Urine will be collected through study session II and III. A study session will take place from 8 am till 2 pm.
optional: muscle metabolic profile (according to Cox et. al. 2016] of a muscle biopsy. | This procedure takes 30 minutes each time and will be performed prior to and immediately post-exercise during study session II and III.
  optional, on a patient-voluntary basis. If consent has been given a total of 4 muscle biopsies will be performed.
optional: individual phenotypic muscle properties (fiber type, mitochondrial density, capillary density | This procedure takes 30 minutes each time and will be performed prior to and immediately post-exercise during study session II and III.
  optional, on a patient-voluntary basis. If consent has been given a total of 4 muscle biopsies will be performed.
Individual physical performance during exercise; VO2 and VCO2 dynamics. | During session I; the maximum exercise test of approximately 12 minutes and during the exercise tests of 15 minutes outside the MR scanner at session II and III.

CONTACTS AND LOCATIONS:
Overall Officials: T.G.J. Derks, MD PhD, Principal Investigator — University Medical Center Groningen
Locations (1):
- University of Groningen, UMC Groningen, Groningen, Netherlands

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Cox PJ, Kirk T, Ashmore T, Willerton K, Evans R, Smith A, Murray AJ, Stubbs B, West J, McLure SW, King MT, Dodd MS, Holloway C, Neubauer S, Drawer S, Veech RL, Griffin JL, Clarke K. Nutritional Ketosis Alters Fuel Preference and Thereby Endurance Performance in Athletes. Cell Metab. 2016 Aug 9;24(2):256-68. doi: 10.1016/j.cmet.2016.07.010. Epub 2016 Jul 27. PMID 27475046
- [Background] Diekman EF, Visser G, Schmitz JP, Nievelstein RA, de Sain-van der Velden M, Wardrop M, Van der Pol WL, Houten SM, van Riel NA, Takken T, Jeneson JA. Altered Energetics of Exercise Explain Risk of Rhabdomyolysis in Very Long-Chain Acyl-CoA Dehydrogenase Deficiency. PLoS One. 2016 Feb 16;11(2):e0147818. doi: 10.1371/journal.pone.0147818. eCollection 2016. PMID 26881790
- [Background] Sentner CP, Hoogeveen IJ, Weinstein DA, Santer R, Murphy E, McKiernan PJ, Steuerwald U, Beauchamp NJ, Taybert J, Laforet P, Petit FM, Hubert A, Labrune P, Smit GPA, Derks TGJ. Glycogen storage disease type III: diagnosis, genotype, management, clinical course and outcome. J Inherit Metab Dis. 2016 Sep;39(5):697-704. doi: 10.1007/s10545-016-9932-2. Epub 2016 Apr 22. PMID 27106217
- [Background] Verbeek RJ, Sentner CP, Smit GP, Maurits NM, Derks TG, van der Hoeven JH, Sival DA. Muscle Ultrasound in Patients with Glycogen Storage Disease Types I and III. Ultrasound Med Biol. 2016 Jan;42(1):133-42. doi: 10.1016/j.ultrasmedbio.2015.08.013. Epub 2015 Oct 3. PMID 26437929
- [Background] Preisler N, Laforet P, Madsen KL, Prahm KP, Hedermann G, Vissing CR, Galbo H, Vissing J. Skeletal muscle metabolism is impaired during exercise in glycogen storage disease type III. Neurology. 2015 Apr 28;84(17):1767-71. doi: 10.1212/WNL.0000000000001518. Epub 2015 Apr 1. PMID 25832663
- [Derived] Hoogeveen IJ, de Boer F, Boonstra WF, van der Schaaf CJ, Steuerwald U, Sibeijn-Kuiper AJ, Vegter RJK, van der Hoeven JH, Heiner-Fokkema MR, Clarke KC, Cox PJ, Derks TGJ, Jeneson JAL. Effects of acute nutritional ketosis during exercise in adults with glycogen storage disease type IIIa are phenotype-specific: An investigator-initiated, randomized, crossover study. J Inherit Metab Dis. 2021 Jan;44(1):226-239. doi: 10.1002/jimd.12302. Epub 2020 Sep 7. PMID 33448466